CLINICAL TRIAL: NCT00052026
Title: A Multicenter, Placebo-Controlled, 8-Month Study of the Effect of Twice Daily Carvedilol in Children With Congestive Heart Failure Due to Systemic Ventricular Systolic Dysfunction
Brief Title: Safety and Efficacy Study of Carvedilol to Treat Children With Congestive Heart Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shaddy, Robert, M.D. (Individual)
Collaborators: University of Utah (Other)
Responsible Party: Robert E Shaddy, MD, The Children's Hospital of Philadelphia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB 105517-321
Record Dates: First submitted 2003-01-21; First posted 2003-01-23 (Estimated); Last update posted 2008-12-25 (Estimated); Status verified 2008-12

CONDITIONS: Congestive Heart Failure
Keywords: Adolescent; Adrenergic alpha-Antagonists/therapeutic use; Adrenergic alpha-Antagonists/pharmacokinetics; Adrenergic alpha-Antagonists/administration & dosage; Adrenergic beta-Antagonists/therapeutic use; Adrenergic beta-Antagonists/pharmacokinetics; Adrenergic beta-Antagonists/administration & dosage; Age Factors; Carbazoles/therapeutic use; Carbazoles/administration & dosage; Child; Child, Preschool; Drug Administration Schedule; Female; Heart Failure, Congestive/etiology; Heart Failure, Congestive/drug therapy; Heart Failure, Congestive/blood; Human; Infant; Infant, Newborn; Male; Natriuretic Peptide, Brain/blood; Placebos; Propanolamines/therapeutic use; Propanolamines/administration & dosage; Prospective Studies; Support, Non-U.S. Gov't; Treatment Outcome; Ventricular Dysfunction/drug therapy; Ventricular Dysfunction/complications; Ventricular Dysfunction/blood; Ventricular Function/drug effects; Ventricular Remodeling/drug effects
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction | interventions — Carvedilol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: placebo
- 2 (Experimental): Low-dose carvedilol
  Interventions: Drug: carvedilol
- 3 (Experimental): high-dose carvedilol
  Interventions: Drug: carvedilol

INTERVENTIONS:
Drug: carvedilol — low-dose carvedilol administered twice daily for 8 months
  Other Names: Coreg
  Arms: 2
Drug: placebo — administered twice daily for 8 months
  Arms: 1
Drug: carvedilol — high-dose carvedilol administered twice daily for 8 months
  Other Names: Coreg
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether a new medicine, called carvedilol, improves symptoms and heart function in children who have congestive heart failure (diminished function of their heart muscle that pumps blood to the body). To accomplish this, we will give carvedilol to some patients who have diminished heart function and congestive heart failure and see whether symptoms and heart function are better at the end of an 8 month period in those who received carvedilol compared to the other patients who did not receive carvedilol. We will be testing 2 different doses of carvedilol compared to no additional medicine.

DETAILED DESCRIPTION:
Overactivity of the sympathetic nervous system is thought to contribute to the pathophysiology of congestive heart failure (CHF). Blockade of the sympathetic nervous system with β-adrenergic inhibitors could be expected to ameliorate these detrimental effects in a manner analogous to the effects of the angiotensin converting enzyme inhibitors on the overactive renin-angiotensin system.

Carvedilol may be superior to pure beta-blockers in the treatment of CHF through its mechanism of action of blocking not only β-receptors but also α-receptors, which would allow vasodilation to reduce the afterload on the failing heart. Since beta-blockers may initially produce a negative inotropic effect on the heart, long term treatment has been needed to show benefits of removal of the adrenergic stimulation. The investigators will monitor the safety and efficacy of carvedilol administration in children with chronic CHF due to systemic ventricular dysfunction.

ELIGIBILITY:
INCLUSION CRITERIA

1. Male or female children from birth through 17 years of age with chronic symptomatic CHF due to systemic ventricular systolic dysfunction who are receiving standard heart failure therapy will be eligible. Since adolescents with left ventricular dysfunction are very similar to adults with this disease, this study will focus recruitment in the prepubertal age group of children, including children from birth through Tanner Stage 3. The number of adolescents enrolled will be limited to approximately 10% of study enrollment. However, teenagers with single ventricles or morphologic right ventricles as systemic ventricles represent an important population that is unique to pediatric cardiology. The 10% limitation will only apply to teenagers who have dilated cardiomyopathies since these patients may be similar to young adults with dilated cardiomyopathies. Adolescents will be defined as Tanner Stage 4 through age 17.
2. A diagnosis of CHF by NYHA Class II-IV (generally, children older than 5 years of age) or Ross' classification of CHF Class II-IV (12) (generally, children less than 5 years old) for at least 1 month (at least 2 weeks, for neonates) prior to screening.
3. An estimated ejection fraction less than 40% in patients with systemic left ventricular dysfunction or qualitative evidence of a dilated ventricle with moderate systemic ventricular systolic dysfunction in patients with right ventricular or single ventricular physiology, documented within 4 weeks of randomization. Patients may be enrolled based on these criteria as determined by the site. However, all echocardiograms will be reviewed and interpreted by the Data Coordinating Center (DCC) at the University of Utah. Upon subsequent review by the DCC, if it is determined that either the ejection fraction is greater than or equal to 40% or the ventricular function is not moderate to severely decreased, patients will be enrolled. However, their data analysis will be based upon the findings from the DCC at the University of Utah.
4. The etiology of the cardiomyopathy will include idiopathic dilated cardiomyopathy, post-viral myocarditis cardiomyopathy, anthracycline-induced cardiomyopathy, ischemic cardiomyopathies (e.g., Kawasaki's disease, repaired anomalous left coronary artery arising from the pulmonary artery, d-TGA s/p arterial switch), cardiomyopathies associated with single ventricle with ventricular systolic dysfunction, corrected transposition, etc. Excluded from enrollment will be dilated cardiomyopathies secondary to muscular dystrophies, hemoglobinopathies, HIV, carnitine deficiency, and systemic ventricular dysfunction due to ventricular outflow obstruction.
5. Patients undergoing treatment for CHF with standard CHF therapy, such as diuretic, digoxin and ACE inhibitors. All patients should be receiving ACE inhibitors prior to enrollment in this study unless contraindicated or intolerant. If intolerance has been established, the patient must have been withdrawn from these drugs for at least one month prior to randomization. Other medications such as hydralazine, nitrates or amiodarone may also be used. Therapy with amiodarone should not have started or stopped within 2 months of randomization.
6. All patients should be receiving diuretics prior to enrollment in this study unless contraindicated or intolerant. Patients must be in optimal fluid status prior to enrollment.
7. Patients must be receiving a stable regimen of standard CHF medications for a period of at least one month (2 weeks in neonates) at the time of randomization into the study.

EXCLUSION CRITERIA

Patients with any of the following will be excluded from the study:

1. NYHA or Ross' CHF Classification Class I (asymptomatic).
2. Patients actively listed for transplantation at time of entry into the study or anticipated to undergo heart transplantation or corrective heart surgery during the 8 months following entry into the study. However, those patients in whom listing for transplantation is anticipated but may be waiting a long period of time (greater than 8 months), such as Status 2 patients, may be considered for enrollment in this study.
3. Sustained or symptomatic ventricular dysrhythmias uncontrolled by drug therapy or the use of an implantable defibrillator, and/or significant cardiac conduction defects, e.g., 2nd degree or 3rd degree AV block, or sick sinus syndrome, unless a functioning pacemaker is in place.
4. Uncorrected primary obstructive or severe regurgitative valvular disease, nondilated (restrictive) or hypertrophic cardiomyopathy, or significant systemic ventricular outflow obstruction.
5. Dilated cardiomyopathies secondary to muscular dystrophies, hemoglobinopathies, HIV, carnitine deficiency, and systemic ventricular dysfunction due to ventricular outflow obstruction.
6. Active myocarditis.
7. Unacceptable blood pressures and heart rates. Sitting (supine in infants) systolic blood pressure must be > 85 mm Hg in teens, > 75 mm Hg in school-aged children, and > 65 mm Hg in infants (12). Resting heart rate must be greater than the 2nd percentile for age (13).
8. Renovascular hypertension or evidence of pulmonary hypertension (pulmonary vascular resistance index > 6 Wood units-m2) unresponsive to vasodilator agents such as oxygen, nitroprusside, or nitric oxide.
9. History or current clinical evidence of moderate-to-severe obstructive pulmonary disease or reactive airway diseases (e.g., asthma) requiring therapy.
10. Significant renal (serum creatinine >2.0), hepatic (serum AST and/or ALT > 3 times upper limit of normal), gastrointestinal, or biliary disorders that could impair absorption, metabolism, or excretion of orally administered medications.
11. Concurrent terminal illness or other severe disease (e.g., active neoplasm) or other significant laboratory value(s) which, in the opinion of the investigator, could preclude participation or survival.
12. Endocrine disorders such as primary aldosteronism, pheochromocytoma, hyper- or hypothyroidism, insulin-dependent diabetes mellitus.
13. Unwillingness or inability to cooperate, or for the parents or guardians to give consent, or for the child to give assent, or any condition of sufficient severity to impair cooperation in the study.
14. Girls of child bearing potential who are pregnant, lactating, or sexually active and not taking adequate contraceptive precautions (e.g., IUD or oral contraceptives for 3 months prior to entry into the study).
15. Use of an investigational drug within 30 days of randomization, or within 5 half-lives of the investigational drug (the longer period will apply); investigational vaccines or biological agents (e.g., the monoclonal antibody Synagis), may be granted exceptions through consultation with the principal investigator and GlaxoSmithKline.
16. History of drug sensitivity or allergic reaction to a-blockers or ß-blockers.
17. Use of any of the following medications within two weeks of randomization:

    * Monoamine oxidase (MAO) inhibitors
    * Calcium entry blockers
    * Alpha blockers, or labetalol
    * Disopyramide, flecainide, encainide, moricizine, propafenone
    * Intravenous ß-adrenergic agonists (including intravenous inotropes such as dobutamine) or intravenous vasodilator agents such as amrinone or milrinone
    * Intravenous CHF medications (e.g., diuretics, digoxin)
18. Treatment with b-adrenergic blockers, including sotalol or carvedilol within 2 months of randomization.

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 161 (Actual)
Dates: Start 2000-05; Primary Completion 2005-06 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is a CHF composite response. | 8 months

SECONDARY OUTCOMES:
Selected individual components of the CHF composite of clinical outcomes | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert E. Shaddy, MD, Principal Investigator — University of Utah
Locations (21):
- United States (21):
  - University of Alabama, Birmingham, Alabama
  - Mattel Children's Hospital at UCLA, Los Angeles, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of Colorado, Denver, Colorado
  - University of Miami, Miami, Florida
  - University of Southern Florida, St. Petersburg, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - Children's Hospital, Boston, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - NYU Medical Center, New York, New York
  - Columbia University, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Childrens Hospital and Regional Medical Center, Seattle, Washington

REFERENCES:
- [Background] Shaddy RE, Curtin EL, Sower B, Tani LY, Burr J, LaSalle B, Boucek MM, Mahony L, Hsu DT, Pahl E, Burch GH, Schlencker-Herceg R. The Pediatric Randomized Carvedilol Trial in Children with Heart Failure: rationale and design. Am Heart J. 2002 Sep;144(3):383-9. doi: 10.1067/mhj.2002.124402. PMID 12228773
- [Background] Boucek MM, Novick RJ, Bennett LE, Fiol B, Keck BM, Hosenpud JD. The Registry of the International Society of Heart and Lung Transplantation: first official pediatric report--1997. J Heart Lung Transplant. 1997 Dec;16(12):1189-206. No abstract available. PMID 9436131
- [Background] Gilbert EM, Anderson JL, Deitchman D, Yanowitz FG, O'Connell JB, Renlund DG, Bartholomew M, Mealey PC, Larrabee P, Bristow MR. Long-term beta-blocker vasodilator therapy improves cardiac function in idiopathic dilated cardiomyopathy: a double-blind, randomized study of bucindolol versus placebo. Am J Med. 1990 Mar;88(3):223-9. doi: 10.1016/0002-9343(90)90146-5. PMID 1968710
- [Background] Waagstein F, Bristow MR, Swedberg K, Camerini F, Fowler MB, Silver MA, Gilbert EM, Johnson MR, Goss FG, Hjalmarson A. Beneficial effects of metoprolol in idiopathic dilated cardiomyopathy. Metoprolol in Dilated Cardiomyopathy (MDC) Trial Study Group. Lancet. 1993 Dec 11;342(8885):1441-6. doi: 10.1016/0140-6736(93)92930-r. PMID 7902479
- [Background] Shaddy RE, Olsen SL, Bristow MR, Taylor DO, Bullock EA, Tani LY, Renlund DG. Efficacy and safety of metoprolol in the treatment of doxorubicin-induced cardiomyopathy in pediatric patients. Am Heart J. 1995 Jan;129(1):197-9. doi: 10.1016/0002-8703(95)90061-6. No abstract available. PMID 7817916
- [Background] Shaddy RE. Beta-blocker therapy in young children with congestive heart failure under consideration for heart transplantation. Am Heart J. 1998 Jul;136(1):19-21. doi: 10.1016/s0002-8703(98)70176-0. PMID 9665213
- [Background] Shaddy RE, Tani LY, Gidding SS, Pahl E, Orsmond GS, Gilbert EM, Lemes V. Beta-blocker treatment of dilated cardiomyopathy with congestive heart failure in children: a multi-institutional experience. J Heart Lung Transplant. 1999 Mar;18(3):269-74. doi: 10.1016/s1053-2498(98)00030-8. PMID 10328154
- [Background] Packer M, Bristow MR, Cohn JN, Colucci WS, Fowler MB, Gilbert EM, Shusterman NH. The effect of carvedilol on morbidity and mortality in patients with chronic heart failure. U.S. Carvedilol Heart Failure Study Group. N Engl J Med. 1996 May 23;334(21):1349-55. doi: 10.1056/NEJM199605233342101. PMID 8614419
- [Background] Bristow MR, Gilbert EM, Abraham WT, Adams KF, Fowler MB, Hershberger RE, Kubo SH, Narahara KA, Ingersoll H, Krueger S, Young S, Shusterman N. Carvedilol produces dose-related improvements in left ventricular function and survival in subjects with chronic heart failure. MOCHA Investigators. Circulation. 1996 Dec 1;94(11):2807-16. doi: 10.1161/01.cir.94.11.2807. PMID 8941106
- [Background] Olsen SL, Gilbert EM, Renlund DG, Taylor DO, Yanowitz FD, Bristow MR. Carvedilol improves left ventricular function and symptoms in chronic heart failure: a double-blind randomized study. J Am Coll Cardiol. 1995 May;25(6):1225-31. doi: 10.1016/0735-1097(95)00012-S. PMID 7722114
- [Background] Richards AM, Doughty R, Nicholls MG, Macmahon S, Ikram H, Sharpe N, Espiner EA, Frampton C, Yandle TG. Neurohumoral prediction of benefit from carvedilol in ischemic left ventricular dysfunction. Australia-New Zealand Heart Failure Group. Circulation. 1999 Feb 16;99(6):786-92. doi: 10.1161/01.cir.99.6.786. PMID 9989964
- [Background] Ross RD, Daniels SR, Schwartz DC, Hannon DW, Shukla R, Kaplan S. Plasma norepinephrine levels in infants and children with congestive heart failure. Am J Cardiol. 1987 Apr 1;59(8):911-4. doi: 10.1016/0002-9149(87)91118-0. PMID 3825955
- [Background] Bristow MR, O'Connell JB, Gilbert EM, French WJ, Leatherman G, Kantrowitz NE, Orie J, Smucker ML, Marshall G, Kelly P, et al. Dose-response of chronic beta-blocker treatment in heart failure from either idiopathic dilated or ischemic cardiomyopathy. Bucindolol Investigators. Circulation. 1994 Apr;89(4):1632-42. doi: 10.1161/01.cir.89.4.1632. PMID 7908610
- [Background] From Nadas AS, Fyler DC: Pediatric Cardiology. 3rd Ed. WB Saunders, Philadelphia, 1972.
- [Background] From Harriet Lane Handbook, 14th Edition, page 132.
- [Derived] Shaddy RE, Boucek MM, Hsu DT, Boucek RJ, Canter CE, Mahony L, Ross RD, Pahl E, Blume ED, Dodd DA, Rosenthal DN, Burr J, LaSalle B, Holubkov R, Lukas MA, Tani LY; Pediatric Carvedilol Study Group. Carvedilol for children and adolescents with heart failure: a randomized controlled trial. JAMA. 2007 Sep 12;298(10):1171-9. doi: 10.1001/jama.298.10.1171. PMID 17848651